CLINICAL TRIAL: NCT01726855
Title: Prevention of Adhesions Following Flexor Tendon Injury Within Zone II With Vascularized Finger Dorsal Fascial Flap
Status: Completed | Type: Observational
Sponsor: The Second Hospital of Tangshan (Other)
Responsible Party: Sponsor
Other Study IDs: sun_rising
Record Dates: First submitted 2012-11-11; First posted 2012-11-15 (Estimated); Last update posted 2024-01-22 (Actual); Status verified 2012-11

CONDITIONS: Tendon Injuries
Keywords: tendon repair
MeSH Terms: conditions — Tendon Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- dorsal fascial flap: combined with standard modified Kessler technique and vascularized finger dorsal fascial flap pedicled with dorsal cutaneous branch of proper digital artery ,which is transported to finger palmar for placement of a mechanical barrier between flexor digitorum superficialis /profundus tendons.
  Interventions: Procedure: vascularized finger dorsal fascial flap
- standard modified Kessler technique

INTERVENTIONS:
Procedure: vascularized finger dorsal fascial flap
  Groups: dorsal fascial flap

SUMMARY:
The purpose of this study was to report a new method of flexor tendon repair in zone II with combined standard modified Kessler technique and vascularized finger dorsal fascial flap pedicled with dorsal cutaneous branch of proper digital artery ,which is transported to finger volar for placement of a mechanical barrier between flexor digitorum superficialis /profundus tendons. The function outcomes of 14 patients (Group A) with flexor tendon repair in zone II with this new technique were compared with those of 32 patients (Group B) with flexor tendon repair in zone II with standard modified Kessler technique. This new technique may prevent serious adhesions between flexor digitorum superficialis /profundus tendons.

ELIGIBILITY:
Inclusion Criteria:

* patients requiring flexor tendon repair or reconstruction within zoneⅡ

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients requiring flexor tendon repair or reconstruction within zoneⅡ
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
the modified Strickland system | 3~12 months
degrees of the maximum active flexion at the distal interphalangeal joint | 3~12 months

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Hospital of Tangshan, Tangshan, Hebei, China